CLINICAL TRIAL: NCT06022094
Title: Effect of a Two-month Carbohydrate-restricted Diet on Energy Metabolism in a Seniors' Residence: The SAGE Study
Brief Title: Effect of a Two-month Carbohydrate-restricted Diet on Energy Metabolism in a Seniors' Residence
Acronym: SAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-5195
Record Dates: First submitted 2023-07-18; First posted 2023-09-01 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Healthy Aging
Keywords: Nutritional intervention; Glucose monitoring; Reduced carb diet; Energy metabolism; Ketones
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Intervention Model Description: All participants will eat a reduced carb menu for 2 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Delta of before/after the intervention (Experimental): Data will be collected before and after the reduced carb intervention
  Interventions: Other: 2 months of reduced carb menus

INTERVENTIONS:
Other: 2 months of reduced carb menus — Participants will eat a reduced carb menu for 2 months
  Other Names: R-CHO

SUMMARY:
The present study will assess the effects on glucose, ketones and other blood biomarkers fuels, cognition, quality of life, physical activity and well-being of a reduced carbohydrate menu (R-CHO) for 2 months in a population living in a residence for the elderly. This intervention study, identified as the SAGE project (phase 2), follows on from the Ketohome project (phase 1) assessing the feasibility of such a project.

DETAILED DESCRIPTION:
Finding an effective therapeutic strategy for Alzheimer's disease (AD) is a societal priority, but it also remains a major challenge. With one exception in 2021, no new pharmaceutical treatment for AD has been approved for over 20 years. However, several clinical trials demonstrate the potential of ketogenic interventions to restore brain energy and improve cognition in people with mild cognitive impairment and AD. Recently, the largest and longest clinical trial of its kind shows that compensating for energy deficit in the brain during aging improves brain metabolic and cognitive functioning in people with early AD and could potentially delay AD.

One of the main types of ketogenic intervention is the highly reduced carbohydrate (5-10% of daily energy value compared to a normal value of 50-65%) and very high fat ketogenic diet. Despite the now well-established safety of the ketogenic diet and its therapeutic value in the treatment of epilepsy and type 2 diabetes, the latter remains difficult to implement in because of the compliance challenge. A reduced glycemic load diet where intake of refined carbohydrates and added sugar is restricted is found to be much less restrictive than a ketogenic diet. Phase 1 of this project showed that decreased carbohydrate (sugar) intake may improve long-term glycemic control and compliance compared to more severe carbohydrate restriction. Having better blood glucose control may also be important in decreasing the risk of AD possibly by improving the metabolic profile and/or by promoting the production and use of ketones. However, its effectiveness in helping cognition in the elderly is still unknown and any changes in dietary habits can be addressed with some resistance.

The objective of this project is therefore to answer the following question: does a reduction in carbohydrates of 30 to 50% for 2 months reduce the risk of AD by improving the metabolic profile in people living in a senior residence?

ELIGIBILITY:
Inclusion Criteria:

* Senior men or women residing in VÜ resident home;
* Understand, read and write French;
* Possess sufficient visual and auditory acuity to pass the cognitive tests;
* Available during the intervention period

Exclusion Criteria:

* Body mass index < 20;
* T1 diabetic;
* Insulin-dependent T2 diabetic;
* Mini Mental State Exam (MMSE) < 20;
* Weight loss >10% in the last 6 months, involuntary or voluntary;
* Known and uncontrolled hypoglycaemia;
* Moderate to severe digestive illnesses that may be aggravated by dietary changes;
* Severe dysphagia;
* Supplementation with medium chain triglycerides oil, ketone salts, ketone ester, adherence to the ketogenic diet, reduced carbohydrate diet, intermittent fasting, or other diet or supplements that may significantly increase ketones in the past month;
* Participation in other intervention research projects on nutrition or aimed at metabolic change simultaneously.
* Medical condition that could prevent the participant from completing the study according to the doctor's opinion

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose levels | 2 months
  Blood glucose will be monitored continuously with a real-time continuous glucose monitor (CGM) for two 10-days periods; before/after intervention in people in a senior residence.
Change in blood ketones levels | 2 months
  Blood ketones will be measured before/after the intervention in people in a senior residence via blood sampling.
Change in blood insulin levels | 2 months
  Blood insulin will be measured before/after the intervention in people in a senior residence via blood sampling.

SECONDARY OUTCOMES:
Change in blood triglycerides levels, | 2 months
  Blood triglycerides levels will be measured before/after the intervention in people in a senior residence via blood sampling.
Change in blood cholesterol levels | 2 months
  Blood cholesterol levels will be measured before/after the intervention in people in a senior residence via blood sampling.
Change in blood glycated hemoglobin levels | 2 months
  Blood glycated hemoglobin levels will be measured before/after the intervention in people in a senior residence via blood sampling.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center on Aging, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vandenberghe C, Hardy E, Morin MC, St-Pierre V, Groulx K, Fortier M, Tessier D, Leclerc P, Cunnane SC. A reduced carbohydrate diet improves glycemic regulation in hyperglycemic older people in a retirement home: the SAGE study. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-10. doi: 10.1139/apnm-2024-0277. Epub 2024 Oct 4. PMID 39366004